CLINICAL TRIAL: NCT05438329
Title: A Phase 1/2a, Multicenter, Open-Label, First in Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of DB-1305 in Subjects With Advanced/Metastatic Solid Tumors
Brief Title: First-in-human Study of DB-1305/BNT325 for Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB-1305-O-1001
Record Dates: First submitted 2022-06-14; First posted 2022-06-29 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (30):
- DB-1305/BNT325 Dose Level 1 (Experimental): Enrolled subjects will receive DB-1305/BNT325 at Dose Level 1
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Level 2 (Experimental): Enrolled subjects will receive DB-1305/BNT325 at Dose Level 2
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Level 3 (Experimental): Enrolled subjects will receive DB-1305/BNT325 at Dose Level 3
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Level 4 (Experimental): Enrolled subjects will receive DB-1305/BNT325 at Dose Level 4
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Level 5 (Experimental): Enrolled subjects will receive DB-1305/BNT325 at Dose Level 5
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Level 6 (Experimental): Enrolled subjects will receive DB-1305/BNT325 at Dose Level 6
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Level 7 (Experimental): Enrolled subjects will receive DB-1305/BNT325 at Dose Level 7
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 in combination with pembrolizumab (Experimental): Enrolled subjects will receive DB-1305/BNT325 in combination with pembrolizumab
  Interventions: Drug: DB-1305/BNT325; Combination Product: Pembrolizumab
- DB-1305/BNT325 Dose Expansion 1 (Experimental): subjects with Non-Small Cell Lung Cancer (NSCLC) with actionable genetic alterations (AGAs) who will receive DB-1305/BNT325 on either dose level 1 or dose level 2
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion 2 (Experimental): Enrolled subjects with NSCLC without AGAs who will receive DB-1305/BNT325 on either dose level 1 or dose level 2
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion 3 (Experimental): Enrolled subjects with OC who will receive DB-1305/BNT325 on either dose level 1 or dose level 2
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion 4 (Experimental): Enrolled subjects with BC who will receive DB-1305/BNT325 on a selected dose level (RP2D)
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion 5 (Experimental): Enrolled subjects with Triple-Negative Breast Cancer (TNBC) who have progressed on or after standard systemic treatments and without prior treatment of sacituzumab govitecan who will receive DB-1305/BNT325 on a selected dose level (RP2D)
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion 6 (Experimental): Enrolled subjects with TNBC with treatment failure on sacituzumab govitecan who will receive DB-1305/BNT325 on a selected dose level (RP2D)
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion 7 (Experimental): Enrolled subjects with EC who will receive DB-1305/BNT325 on a selected dose level (RP2D)
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion 8 (Experimental): Enrolled subjects with malignant mesothelioma will receive DB-1305/BNT325 on a selected dose level (RP2D)
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion 9 (Experimental): Enrolled subjects with Cervical Cancer (CC) who will receive DB-1305/BNT325 on a selected dose level (RP2D)
  Interventions: Drug: DB-1305/BNT325
- Experimental: DB-1305/BNT325 Dose Expansion 10 (Experimental): Enrolled subjects with pancreatic cancer who will receive DB-1305/BNT325 on a selected dose level (RP2D)
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion 11 (Experimental): Enrolled subjects with Castration-Resistant Prostate Cancer (CRPC) who will receive DB-1305/BNT325 on a selected dose level (RP2D)
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion PB1 (Experimental): Enrolled subjects with NSCLC without AGAs who will receive DB-1305/BNT325 on a selected dose level in combination with pembrolizumab
  Interventions: Drug: DB-1305/BNT325; Combination Product: Pembrolizumab
- Experimental: DB-1305/BNT325 Dose Level 8 (Experimental): Enrolled subjects will receive DB-1305/BNT325 at Dose Level 8
  Interventions: Drug: DB-1305/BNT325
- Experimental: DB-1305/BNT325 in combination with BNT327 (Experimental): Enrolled subjects will receive DB-1305/BNT325 in combination with BNT327
  Interventions: Drug: DB-1305/BNT325; Drug: BNT327
- Experimental: DB-1305/BNT325 Dose Expansion PM1 (Experimental): Enrolled subjects with NSCLC without AGAs who will receive DB-1305/BNT325 on a selected dose level in combination with BNT327
  Interventions: Drug: DB-1305/BNT325; Drug: BNT327
- Experimental: DB-1305/BNT325 Dose Expansion PM2 (Experimental): Enrolled subjects with NSCLC with AGAs who will receive DB-1305/BNT325 on a selected dose level in combination with BNT327
  Interventions: Drug: DB-1305/BNT325; Drug: BNT327
- Experimental: DB-1305/BNT325 Dose Expansion PM3 (Experimental): Enrolled subjects with CC who will receive DB-1305/BNT325 on a selected dose level in combination with BNT327
  Interventions: Drug: DB-1305/BNT325; Drug: BNT327
- Experimental: DB-1305/BNT325 Dose Expansion PM4 (Experimental): Enrolled subjects with OC who will receive DB-1305/BNT325 on a selected dose level in combination with BNT327
  Interventions: Drug: DB-1305/BNT325; Drug: BNT327
- Experimental: DB-1305/BNT325 Dose Expansion PM5 (Experimental): Enrolled subjects with TNBC who will receive DB-1305/BNT325 on a selected dose level in combination with BNT327
  Interventions: Drug: DB-1305/BNT325; Drug: BNT327
- DB-1305/BNT325 Dose Expansion 12 (Experimental): Enrolled subjects with head and neck cancer who will receive DB-1305/BNT325 on a selected dose level (RP2D)
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Level 9 (Experimental): Enrolled subjects will receive DB-1305/BNT325 at Dose Level 9
  Interventions: Drug: DB-1305/BNT325
- DB-1305/BNT325 Dose Expansion PM6 (Experimental): Enrolled subjects with NSCLC without AGA who will receive DB-1305/BNT325 on a selected dose level in combination with BNT327
  Interventions: Drug: DB-1305/BNT325; Drug: BNT327

INTERVENTIONS:
Drug: DB-1305/BNT325 — Administered Injection of Vein (I.V.)
  Other Names: DB-1305/BNT325 for Injection
Combination Product: Pembrolizumab — Administered I.V.
  Arms: DB-1305/BNT325 Dose Expansion PB1; DB-1305/BNT325 in combination with pembrolizumab
Drug: BNT327 — Administered I.V.
  Arms: DB-1305/BNT325 Dose Expansion PM6; Experimental: DB-1305/BNT325 Dose Expansion PM1; Experimental: DB-1305/BNT325 Dose Expansion PM2; Experimental: DB-1305/BNT325 Dose Expansion PM3; Experimental: DB-1305/BNT325 Dose Expansion PM4; Experimental: DB-1305/BNT325 Dose Expansion PM5; Experimental: DB-1305/BNT325 in combination with BNT327

SUMMARY:
This is a dose-escalation and dose-expansion Phase 1/2a trial to evaluate the safety and tolerability of DB-1305/BNT325 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, multiple-dose, first in human (FIH) study. The study consists of two parts: Part 1 adopts an accelerated titration at first dose level followed with classic "3+3" design to identify the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D); Part 2 is a dose expansion phase to confirm the safety, tolerability and explore efficacy in selected malignant solid tumors at the MTD/the RP2D. This study will enroll subjects with advanced/unresectable, recurrent, or metastatic malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (defined as ≥ 18 years of age or acceptable age according to local regulations at the time of voluntarily signing of informed consent).
* Histologically or cytologically confirmed unresectable advanced/ metastatic solid tumors who have relapsed or progressed on or after standard systemic treatments or for which no standard treatment is available.
* At least one measurable lesion as assessed by the investigator according to RECIST version 1.1 criteria.
* Has a life expectancy of ≥ 3 months.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
* Has Left Ventricular Ejection Fraction (LVEF) ≥ 50% by either echocardiography (ECHO) or multiple-gated acquisition (MUGA) within 28 days before enrollment.
* Has adequate organ functions within 7 days prior to Day 1 of Cycle 1.
* Has adequate treatment washout period prior to Day 1 of Cycle 1.
* Is willing to provide pre-existing resected tumor samples or undergo fresh tumor biopsy for the measurement of Trop-2 level and other biomarkers if not contraindicated.
* Is capable of comprehending study procedures and risks outlined in the informed consent and able to provide written consent and agree to comply with the requirements of the study and the schedule of assessments.

Exclusion Criteria:

* Has a medical history of symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] classes II-IV) or serious cardiac arrhythmia requiring treatment.
* Has a medical history of myocardial infarction or unstable angina within 6 months before enrollment.
* Has an average of Fredericia's formula-QT corrected interval (QTcF) prolongation to > 470 millisecond (ms) in males and females based on a 12-lead electrocardiogram (ECG) in triplicate.
* Has a medical history of non-infectious Interstitial Lung Diseases (ILD)/pneumonitis or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Has a lung-specific intercurrent clinically significant illness.
* Has an uncontrolled infection requiring IV injection of antibiotics, antivirals, or antifungals.
* Subjects have human immunodeficiency virus (HIV) infection with acquired immune deficiency syndrome (AIDS) defining illness are not eligible for enrollment; However, subjects have had HIV infection with a cluster of differentiation 4 (CD4)+ T cell count > 350 cells/µL and no history of an AIDS-defining illness are eligible for entry.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1123 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of Participants with Dose-Limiting Toxicities (DLTs) as assessed by National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. | up to 21 days after Cycle 1 Day 1
  Percentage of participants in Part 1 with DLTs
Phase 1: Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) as assessed by CTCAE v5.0. | Up to 30 days after last study treatment administration or before starting new anticancer treatment, whichever comes first.
  Percentage of participants with TEAEs in Part 1 graded according to NCI CTCAE v5.0
Phase 1: Percentage of Participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up 30 days after last study treatment administration or before starting new anticancer treatment, whichever comes first.
  Percentage of Participants with SAEs in Part 1 graded according to NCI CTCAE v5.0
Maximum Tolerated Dose (MTD) of DB-1305/BNT325 | At the end of Cycle 1 (each cycle is 21 days)
  MTD on the data collected during Part 1
Phase 1: RP2D of DB-1305/BNT325 | From first study treatment administration until the initiation of Phase 2a, approximately up to 12 months.
  RP2D of DB-1305/BNT325 based on the data collected during Part 1
Phase 2a: Percentage of Participants with TEAEs as assessed by CTCAE v5.0. | Up to 30 days after last study treatment administration or before starting new anticancer treatment, whichever comes first.
  Percentage of participants with TEAEs in Part 2 graded according to NCI CTCAE v5.0 (secondary outcome measure in cohort 3)
Phase 2a: Percentage participants with SAEs as assessed by CTCAE v5.0. | Up to 30 days after last study treatment administration or before starting new anticancer treatment, whichever comes first.
  Percentage of participants with SAEs in Part 2 graded according to NCI CTCAE v5.0 (secondary outcome measure in cohort 3)
Phase 2a: Objective Response Rate (ORR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. | Up to disease progression or death or before starting new anticancer treatment or withdrawal from the trial, whichever comes first, approximately up to 12 months.
  The percentage of subjects who had a best response rating of CR and PR

SECONDARY OUTCOMES:
Phase 1: ORR will be determined from tumor assessments by investigator per RECIST 1.1 | with 8 cycles (each cycle is 21 days)
  Phase 1: ORR will be determined from tumor assessments by investigator per RECIST 1.1
Phase 1 & Phase 2a: duration of response (DoR) will be determined from tumor assessments by investigator per RECIST 1.1 | with 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: duration of response (DoR) will be determined from tumor assessments by investigator (by BICR in cohort 3 in Phase 2a) per RECIST 1.1
Phase 1 & Phase 2a: disease-control rate (DCR) | with 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: disease-control rate (DCR)
Phase 1 & Phase 2a: time to response (TTR) | with 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: time to response (TTR)
Phase 1 & Phase 2a: progression free survival (PFS) will be determined from tumor assessments by investigator per RECIST 1.1 | with 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: progression free survival (PFS) will be determined from tumor assessments by investigator (by BICR in cohort 3 in Phase 2a) per RECIST 1.1
Phase 1 & Phase 2a: overall survival (OS) | with 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: overall survival (OS)
Phase 1 & Phase 2a: Pharmacokinetic parameters: (the area under the concentration-time curve from the time zero to the last quantifiable concentration [AUC0-last] of DB-1305/BNT325 | within 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: Pharmacokinetic parameters: (the area under the concentration-time curve from the time zero to the last quantifiable concentration [AUC0-last] of DB-1305/BNT325
Phase 1 & Phase 2a: Pharmacokinetic parameters: the area under the concentration-time curve from time 0 to tau [AUC0-tau] of DB-1305/BNT325 | within 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: Pharmacokinetic parameters: the area under the concentration-time curve from time 0 to tau [AUC0-tau] of DB-1305/BNT325
Phase 1 & Phase 2a: peak observed concentration [Cmax] of DB-1305/BNT325 | within 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: peak observed concentration [Cmax] of DB-1305/BNT325
Phase 1 & Phase 2a: Pharmacokinetic parameters: time to Cmax [Tmax] of DB-1305/BNT325 | within 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: Pharmacokinetic parameters: time to Cmax [Tmax] of DB-1305/BNT325
Phase 1 & Phase 2a: Pharmacokinetic parameters: trough concentration [Ctrough] of DB-1305/BNT325 | within 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: Pharmacokinetic parameters: trough concentration [Ctrough] of DB-1305/BNT325
Phase 1 & Phase 2a: anti-drug antibody (ADA) prevalence: the proportion of subjects who are ADA positive at any point in time (at baseline and post-baseline). ADA incidence: the proportion of subjects having treatment-emergent ADA. | within 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: anti-drug antibody (ADA) prevalence of DB-1305: the proportion of subjects who are ADA positive at any point in time (at baseline and post-baseline). ADA incidence of DB-1305: the proportion of subjects having treatment-emergent ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hu, Study Director — DualityBio Inc.
Locations (30):
- United States (12):
  - Site 103, Cerritos, California
  - Site 108, Los Angeles, California
  - D&H Cancer Research Center Llc, Margate, Florida
  - Site 109, Plantation, Florida
  - BRCR Medical Center Inc., Tamarac, Florida
  - Site 106, Detroit, Michigan
  - Site 102, New York, New York
  - Site 101, Canton, Ohio
  - Site 105, Nashville, Tennessee
  - Site 110, Arlington, Texas
  - Site 104, Houston, Texas
  - Site 107, Fairfax, Virginia
- China (17):
  - Site 211, Bengbu, Anhui
  - Site 217, Hefei, Anhui
  - Site 213, Fuzhou, Fujian
  - Site 209, Nanning, Guangxi
  - Site 221, Guigang, Guanxi
  - Site 202, Zhengzhou, Henan
  - Site 205, Wuhan, Hubei
  - Site 208, Ganzhou, Jiangxi
  - Site 201, Changchun, Jilin
  - Site 210, Shenyang, Liaoning
  - Site 216, Jinan, Shandong
  - Site 212, Linyi, Shandong
  - Site 207, Shanghai, Shanghai Municipality
  - Site 206, Chengdu, Sichuan
  - Site 203, Tianjin, Tianjin Municipality
  - Site 220, Taizhou, Zhejiang
  - Site 219, Guangzhou
- BRCR GLOBAL Puerto Rico LLC., Mayagüez, Puerto Rico

IPD SHARING:
Plan to Share IPD: No